CLINICAL TRIAL: NCT04749940
Title: PRF Based Dressing Versus AQUACEL® for Local Treatment of Skin Graft Donor Site: A Non-Inferiority Trial
Brief Title: PRF Based Dressing Versus AQUACEL® for Local Treatment of Skin Graft Donor Site
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no bugdet for the study
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Yehuda Ullmann MD, Professor, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0007-21
Record Dates: First submitted 2021-02-01; First posted 2021-02-11 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Treatment of Skin Graft Donor Site
MeSH Terms: interventions — Carboxymethylcellulose Sodium

STUDY DESIGN:
Intervention Model Description: A prospective single-blind study, where the evaluator is blinded to the treatment. Each patient will be dressed with both Aquacel® and PRF dressing. Half of the donor site area will be dressed with PRF dressing, and half with Aquacel®.
Masking Description: Each patient will be dressed with both Aquacel® and PRF dressing. Half of the donor site area will be dressed with PRF dressing, and half with Aquacel®.
  3 days after surgery the patients will be asked to complete a VAS questionnaire. A week and 2 weeks after surgery, patients will have their dressing changed as in the first treatment, and will answer VAS(9) and bluebelle(10) questionnaires. The wound will be photographed again for follow-up. Three weeks, 6 weeks and 3 months after surgery the scar in the donor area will be evaluated. The photographs will be shown to the blinded evaluator, to evaluate wound healing by epithelialization estimation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospitalized burn patients (Experimental): Half of the donor site area will be dressed with PRF dressing, and half with Aquacel®.
  Interventions: Other: Half of the harvested area will be dressed with PRF dressing, and half with Aquacel®.

INTERVENTIONS:
Other: Half of the harvested area will be dressed with PRF dressing, and half with Aquacel®. — Half of the harvested area will be dressed with PRF dressing, and half with Aquacel®.

SUMMARY:
PRF Based Dressing Versus AQUACEL® for Local Treatment of Skin Graft Donor Site: A Non-Inferiority Trial

DETAILED DESCRIPTION:
A prospective single-blind study, where the evaluator is blinded to the treatment. Each patient will be dressed with both Aquacel® and PRF dressing. Half of the donor site area will be dressed with PRF dressing, and half with Aquacel®.

3 days after surgery the patients will be asked to complete a VAS questionnaire. A week and 2 weeks after surgery, patients will have their dressing changed as in the first treatment, and will answer VAS(9) and bluebelle(10) questionnaires. The wound will be photographed again for follow-up. Three weeks, 6 weeks and 3 months after surgery the scar in the donor area will be evaluated. The photographs will be shown to the blinded evaluator, to evaluate wound healing by epithelialization estimation.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a small burn (2-20% TBSA), who require skin grafting.

Exclusion Criteria:

* Patients younger than 18 years
* Patients refusing hospitalization
* Patients with heavily infected wounds, which are the probable cause of bacteremia or sepsis.
* Patients with diabetes mellitus or peripheral vascular disease
* Patients under treatment of steroids or other immunosuppressing agents
* Patients with infectious diseases, i.e., HIV, HCV or HBV.
* Patients who are smokers.
* Patients with a known allergy to the dressing.
* Female patients who are pregnant or nursing, psychiatric patients and soldiers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change of percentage of wound healing after 1 week, 2 weeks and 3 weeks. | 3 weeks
  Primary variables will be analyzed using ImageJ software.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Peck MD. Epidemiology of burns throughout the world. Part I: Distribution and risk factors. Vol. 37, Burns. Burns; 2011. p. 1087-100. 2. Lee RC, Teven CM. Acute Management of Burn/Electrical Injuries. In: Song DH, editor. Neligen's Plastic Surgery. 4th ed. Elsevier Ltd; 2018. p. 391-423. 3. Ding X, Shi L, Liu C, et al. A randomized comparison study of Aquacel Ag and Alginate Silver as skin graft donor site dressings. Burns. 2013 Dec;39(8):1547-50. 4. Haith LR, Stair Buchmann ME, Ackerman BH, et al. Evaluation of Aquacel Ag for Autogenous Skin Donor Sites. J Burn Care Res. . Nov-Dec 2015;36(6):602-6. 5. Sousa F, Machado V, Botelho J, Proença L, Mendes JJ, Alves R. Effect of A-PRF Application on Palatal Wound Healing after Free Gingival Graft Harvesting: A Prospective Randomized Study. Eur J Dent [Internet]. 2020 Feb 1 [cited 2020 Sep 20];14(1):63-9. Available from: https://pubmed.ncbi.nlm.nih.gov/32168533/ 6. Chou TM, Chang HP, Wang JC. Autologous platelet concentrates in maxillofacial regenerative therapy [Internet]. Vol. 36, Kaohsiung Journal of Medical Sciences. John Wiley and Sons Inc.; 2020 [cited 2020 Sep 20]. p. 305-10. Available from: https://pubmed.ncbi.nlm.nih.gov/32052598/ 7. Somani A, Rai R. Comparison of efficacy of autologous platelet-rich fibrin versus saline dressing in chronic venous leg ulcers: A randomised controlled trial. J Cutan Aesthet Surg [Internet]. 2017 Jan 1 [cited 2020 Sep 20];10(1):8-12. Available from: https://pubmed.ncbi.nlm.nih.gov/28529414/ 8. Wang L, Liu G, Li Z, Jia BC, Wang Y. Clinical application of platelet-rich fibrin in chronic wounds combined with subcutaneous stalking sinus. Zhonghua Shao Shang Za Zhi [Internet]. 2018 Sep 20 [cited 2020 Sep 20];34(9):637-42. Available from: https://pubmed.ncbi.nlm.nih.gov/30293368/ 9. Piccin A, Di Pierro AM, Canzian L, Primerano M, Corvetta D, Negri G, et al. Platelet gel: A new therapeutic tool with great potential [Internet]. Vol. 15, Blood Transfusion. SIMTI Servizi Sri; 2017 [cited 2020 Sep 20]. p. 333-40. Available from: https://pubmed.ncbi.nlm.nih.gov/27483482/ 10. Ding Y, Cui L, Zhao Q, et al. Platelet-Rich Fibrin Accelerates Skin Wound Healing in Diabetic Mice. Ann Plast Surg. 2017 Sep;79(3):e15-e19. 11. Yüce E, Kömerik N. Potential effects of advanced platelet rich fibrin as a wound-healing accelerator in the management of alveolar osteitis: A randomized clinical trial. Niger J Clin Pract. 2019 Sep;22(9):1189-1195. 12. Alpan AL, Cin GT. PRF improves wound healing and postoperative discomfort after harvesting subepithelial connective tissue graft from palate: a randomized controlled trial. Clin Oral Investig. 2020 Jan;24(1):425-436. 13. Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis [Internet]. 1978 [cited 2020 Sep 20];37(4):378-81. Available from: https://pubmed.ncbi.nlm.nih.gov/686873/ 14. Macefield R, Blazeby J, Reeves B, Brookes S, Avery K, Rogers C, et al. Validation of the Bluebelle Wound Healing Questionnaire for assessment of surgical-site infection in closed primary wounds after hospital discharge. BJS [Internet]. 2019 Feb 17 [cited 2020 Sep 20];106(3):226-35. Available from: https://onlinelibrary.wiley.com/doi/abs/10.1002/bjs.11008